CLINICAL TRIAL: NCT04757831
Title: A Prospective Study of COVID-19 and Related Outcomes in School Aged Children (ABC Health Outcomes in Children)
Brief Title: Coronavirus-19 (COVID-19) and Related Outcomes in School Aged Children (ABC Health Outcomes in Children)
Status: Withdrawn | Type: Observational
Why Stopped: Study did not begin
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00107647
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-02

CONDITIONS: Covid19; MIS-C
MeSH Terms: conditions — COVID-19; pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational study with a primary objective of determining the incidence of non-severe and severe COVID-19, including MIS-C, among eligible children who are diagnosed with COVID-19 and consent (or assent) to collection of data on risk factors using a unique direct-to-participant, direct-to-family, and direct-to-community approach. Secondary and exploratory objectives include risk factors of severe disease and quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Participant is ≤ 21 years of age at time of enrollment
* Participant or their parent/guardian has downloaded the "ABC Science" App from the App store as a part of the ABC Science Collaborative (Pro00107785) and has agreed to the App's Terms of Use
* Participant has a positive COVID-19 diagnosis, defined as one or more of the following:

  1. A positive COVID-19 test; or
  2. Clinical diagnosis of COVID-19 based on symptoms, as documented by a medical provider, in the absence of a positive influenza test; or
  3. Retrograde diagnosis based on presence of COVID-19 antibodies

Exclusion Criteria:

* N/A

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants ≤ 21 years of age who have a COVID-19 diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Describe the incidence of non-severe and severe COVID-19, including Multisystem Inflammatory Syndrome in Children (MIS-C). | 90 days
  Number of participants who report non-severe or severe COVID-19 disease (defined as a hospitalization event, severe neurological dysfunction, occurrence of MIS-C, or death within 90 days of infection with SARS-CoV-2), reported as a proportion (%) of the total number of participants enrolled in the study who develop non-severe and severe COVID-19 from the time of study initiation to the end of study.

SECONDARY OUTCOMES:
Describe risk factors of non-severe and severe COVID-19. | Up to 5 years
  Demographic variables (e.g. English proficiency, internet access, school district, age, race)
Describe risk factors of non-severe and severe COVID-19. | Up to 5 years
  COVID-19-related symptoms (e.g. cough, fever, shortness of breath, headache, loss of smell)
Describe risk factors of non-severe and severe COVID-19. | Up to 5 years
  Type of COVID-19 exposure (e.g. household, school-related, travel, other, unknown)
Characterize outcomes associated with COVID-19 in children. | Up to 5 years
  Incidence of subsequent exposures to COVID-19 from baseline to the end of study.
Characterize outcomes associated with COVID-19 in children. | Up to 5 years
  Incidence of ongoing COVID-19 symptoms from baseline to the end of study.
Characterize outcomes associated with COVID-19 in children. | Up to 5 years
  Duration of ongoing COVID-19 symptoms from baseline to the end of study.
Characterize outcomes associated with COVID-19 in children. | Up to 5 years
  Incidence of hospitalizations from baseline to the end of study.
Characterize outcomes associated with COVID-19 in children. | Up to 5 years
  Duration of hospitalizations from baseline to the end of study.
Characterize outcomes associated with COVID-19 in children. | Up to 5 years
  Incidence of neurologic complications from baseline to the end of study.
Characterize outcomes associated with COVID-19 in children. | Up to 5 years
  Duration of neurologic complications from baseline to the end of study.
Characterize outcomes associated with COVID-19 in children. | Up to 5 years
  Incidence of COVID-19 vaccination from baseline to the end of study.
Describe characteristics of participants who attend in-person versus virtual classes. | Up to 5 years
  Baseline demographics of those who attend in-person classes compared to those who do not.
Describe the duration of in-person school attendance. | Up to 5 years
  Average in-person attendance from the first day of school to the last day of school among participants compared to the national average during each school year.

CONTACTS AND LOCATIONS:
Overall Officials: Kanecia Zimmerman, MD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This study is a part of the ABC Science Collaborative. — https://abcsciencecollaborative.org/